CLINICAL TRIAL: NCT02934906
Title: A Multi-center Prospective Cohort Study on the Anti-HPA Antibodies Caused Neonatal Alloimmune Thrombocytopenia in Chinese Pregnant Women
Brief Title: Study on the Anti-HPA Antibodies Caused Neonatal Alloimmune Thrombocytopenia in Chinese Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Air Force Military Medical University, China (Other); Shengjing Hospital (Other); Qilu Hospital of Shandong University (Other); Second Xiangya Hospital of Central South University (Other); LanZhou University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Sir Run Run Shaw Hospital (Other); Jilin University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Second Affiliated Hospital of Nanchang University (Other); Guangzhou First People's Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Beijing Chao Yang Hospital (Other); Qingdao University (Other); Peking University First Hospital (Other); RenJi Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); MCH Hospital of Yinchuan City (Unknown); Henan Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Zhongjun Li, Professor, Chief of Blood Transfusion Department, Xinqiao Hospital of Chongqing
Other Study IDs: V2.0(20160720)
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Neonatal Alloimmune Thrombocytopenia
Keywords: Neonatal Alloimmune Thrombocytopenia; pregnancy; human platelet allogantigen; asian; Chinese
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: Pregnant women with anti-HPA antibody negative from the same hospital, the same race, and the same gravidity and parity, who are admitted at the same time.
  Interventions: Procedure: Standard clinical treatment, including intravenous immunoglobulin and/or platelet transfusion
- Experimental Group: pregnant women with anti-HPA antibody positive
  Interventions: Procedure: Standard clinical treatment, including intravenous immunoglobulin and/or platelet transfusion

INTERVENTIONS:
Procedure: Standard clinical treatment, including intravenous immunoglobulin and/or platelet transfusion — Observational study.

SUMMARY:
This clinical study aims to investigate the anti-HPA antibodies caused neonatal alloimmune thrombocytopenia in Chinese pregnant women. The survey and data collect will help form an appropriate clinical screening procedure

ELIGIBILITY:
Inclusion Criteria:

* 12-28 weeks pregnant Chinese women
* between Jan 1, 2017 and Dec 31, 2018

Exclusion Criteria:

* Not willing to participate in this study
* Plan to terminate pregnancy early

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Chinese women and their new borns
Sampling Method: Non-Probability Sample
Enrollment: 55497 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The positive rate of anti-HPA antibody | Up to one and a half years after the study completed
The morbidity of NAIT | Up to one and a half years after the study completed

SECONDARY OUTCOMES:
Antigenic specificity of anti-HPA antibodies | Up to one and a half years after the study completed
Association of anti-HPA antibody with HLA genotype as assessed by Chi-square test | Up to one and a half years after the study completed
The relationship between the titer of anti-HPA antibody and clinical symptom severity in NAIT as assessed by Spearman Correlation assay | Up to one and a half years after the study completed

REFERENCES:
- [Derived] Chen L, Liu Z, Liu T, Ma X, Rao M, Wang Y, Sun B, Yin W, Zhang J, Yan B, Li X, Wang Q, Zhang L, Wen J, Liu F, Wang P, Wei Y, Huang Y, Wu J, Guo Y, Kang Y, Song X, Liu X, Zhang G, Xie T, Chen Y, Zeng X, Li Z. Neonatal alloimmune thrombocytopenia caused by anti-HPA antibodies in pregnant Chinese women: a study protocol for a multicentre, prospective cohort trial. BMC Pregnancy Childbirth. 2017 Aug 31;17(1):281. doi: 10.1186/s12884-017-1453-y. PMID 28859622